CLINICAL TRIAL: NCT04520061
Title: Developing a Health Insurance Navigation Program for Survivors of Childhood Cancer
Acronym: HINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other); St. Jude Children's Research Hospital (Other); University of Utah (Other)
Responsible Party: Principal Investigator, Elyse Park, PhD, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018P003088
Record Dates: First submitted 2020-08-12; First posted 2020-08-20 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Health Insurance; Childhood Cancer Survivors
Keywords: survivorship

STUDY DESIGN:
Intervention Model Description: Intervention; enhanced usual care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigation Intervention (Experimental): The intervention will be delivered via synchronous videoconferencing (real-time delivery and communication between the navigator and the participant) by a trained patient navigator and will consist of 4, 30-minute sessions delivered every week, over the span of one month. The navigation intervention group will also receive a mailed copy of the brochure.
  Interventions: Behavioral: Health Insurance Navigation Program
- Enhanced Usual Care (No Intervention): Enhanced usual care will consist of an online or mailed health insurance resource guide.

INTERVENTIONS:
Behavioral: Health Insurance Navigation Program — The program will be delivered via videoconferencing by a navigator over a 2-month period and will consist of 4 sessions. The navigation intervention sessions will be as follows: Session 1- Learning About Survivorship Healthcare Needs; Session 2- Learning About Your Plan in Relation to Policy; Session 3- Navigating One's Own Plan and Overcoming Obstacles; Session 4- Managing Care Costs.
  Arms: Navigation Intervention

SUMMARY:
Dr. Park and her colleagues published findings in the Journal of Clinical Oncology demonstrating that CCSS survivors, compared to siblings, were significantly more likely to be uninsured and to have difficulties obtaining health insurance. Given the current insurance landscape and the additional insurance burden that childhood cancer survivors face, the present study seeks to develop and pilot a health insurance navigation program targeted at feasibility and acceptability with survivors, and improving health insurance literacy and ameliorating financial distress related to medical costs. The proposed health insurance navigation will involve 4 navigator-led health insurance navigation sessions. The study investigators propose that, compared to the control arm (who will receive a health insurance information guide, but will not receive the navigation intervention), participants in the intervention arm will have improved health insurance literacy and decreased financial distress related to medical costs.

DETAILED DESCRIPTION:
The present study seeks to develop and pilot a health insurance navigation program with childhood cancer survivors recruited from the Long-Term Follow-Up (LTFU) Cohort. Childhood cancer survivors tend to face health challenges throughout their lives that require monitoring and ongoing care. This is compounded by the tendency among childhood survivors to have higher rates of under and uninsurance, unmet healthcare need, and burdensome costs related to care.These burdensome costs also contribute to underutilization of care among survivors. Additionally, as health insurance systems and designs continue to evolve, many people have inadequate understandings of their own health insurance. Dr. Park and her colleagues published findings that suggested LTFU survivors had difficulty in understanding how to use their insurance, and often experienced financial-related distress. Survivors were more likely than their siblings to have borrowed money to pay for medical expenses, and only 27.3% of survivors and 26.2% of their siblings reported familiarity with the ACA. Given these circumstances, understanding and navigating insurance benefits in the current in the current landscape is crucial for cancer survivors to obtain and utilize the health care that they need. With this in mind, the study investigators propose to develop and pilot an insurance navigation intervention with LTFU participants.

The three institutions involved in this study have differing, complementary roles that will contribute to the development and piloting of a health insurance navigation intervention. As the lead site and IRB of record for this study, Massachusetts General Hospital (MGH) will be responsible for the development and regulation of all study-related materials. MGH will also be responsible for the delivery of the navigation intervention (which necessitates the training and supervision of the individual delivery the navigation).

As a collaborating site for this study, St. Jude Children's Research Hospital will be responsible for all recruitment activities, as this study plans to recruit exclusively from the Long-Term Follow-Up Study (LTFU) Cohort.

As a collaborating site for this study, the University of Utah will be responsible for all participant assessment during the study, which will include baseline and follow-up surveys, and exit interviews.

Approximately 80 LTFU participants will be recruited for the randomized pilot trial portion of the study. Prospective participants for the pilot randomized trial portion of the study will be identified via LTFU records, and recruited and consented by LTFU study staff at St. Jude Children's Research Hospital. Prospective participants will receive an invitation to the study through email and mail. The proposed navigation intervention will be delivered by a health insurance navigator via HIPAA-compliant videoconferencing. Content of the navigation intervention will involve the following sessions: 1- Learning Abut Survivorship Healthcare Needs; 2- Learning About Your Plan in Relation to Policy; 3- Navigating One's Own Plan and Overcoming Obstacles; 4- Managing Care Costs. The sessions will be delivered to participants every week over a one to two-month period. Participants will be randomized into either the navigation intervention arm, or the enhanced usual care arm (approximately 40 per arm). The sample size of approximately 40 per arm was chosen to enable evaluation of feasibility and acceptability goals, as well as to explore meaningful differences in the outcomes.To assess the proposed primary and secondary outcomes, all trial participants will complete a baseline and 3-month post-program follow-up survey (approximately 5-month follow-up from baseline). The surveys will be conducted via RedCap or via mailed survey (which will then be input into the RedCap database by study staff). Intervention arm participants will also complete an exit interview in order to further refine the navigation intervention. Both study arm participants will receive a health insurance information guide.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* access to a smartphone, computer, or tablet with internet access
* currently has health insurance

Exclusion Criteria:

* under 18 years of age
* unable to give consent due to psychiatric or cognitive impairment
* lack of access to a smartphone, computer, or tablet with internet access
* does not currently have health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elyse R Park, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
We will not make individual participant data available to any researchers outside of those approved to work on the study under the central IRB.

REFERENCES:
- [Background] Park ER, Li FP, Liu Y, Emmons KM, Ablin A, Robison LL, Mertens AC; Childhood Cancer Survivor Study. Health insurance coverage in survivors of childhood cancer: the Childhood Cancer Survivor Study. J Clin Oncol. 2005 Dec 20;23(36):9187-97. doi: 10.1200/JCO.2005.01.7418. PMID 16361621
- [Background] Robison LL, Hudson MM. Survivors of childhood and adolescent cancer: life-long risks and responsibilities. Nat Rev Cancer. 2014 Jan;14(1):61-70. doi: 10.1038/nrc3634. Epub 2013 Dec 5. PMID 24304873
- [Background] Park ER, Kirchhoff AC, Zallen JP, Weissman JS, Pajolek H, Mertens AC, Armstrong GT, Robison LL, Donelan K, Recklitis CJ, Diller LR, Kuhlthau KA. Childhood Cancer Survivor Study participants' perceptions and knowledge of health insurance coverage: implications for the Affordable Care Act. J Cancer Surviv. 2012 Sep;6(3):251-9. doi: 10.1007/s11764-012-0225-y. Epub 2012 May 17. PMID 22592507
- [Background] Oeffinger KC, Mertens AC, Hudson MM, Gurney JG, Casillas J, Chen H, Whitton J, Yeazel M, Yasui Y, Robison LL. Health care of young adult survivors of childhood cancer: a report from the Childhood Cancer Survivor Study. Ann Fam Med. 2004 Jan-Feb;2(1):61-70. doi: 10.1370/afm.26. PMID 15053285
- [Background] Yeazel MW, Oeffinger KC, Gurney JG, Mertens AC, Hudson MM, Emmons KM, Chen H, Robison LL. The cancer screening practices of adult survivors of childhood cancer: a report from the Childhood Cancer Survivor Study. Cancer. 2004 Feb 1;100(3):631-40. doi: 10.1002/cncr.20008. PMID 14745882
- [Background] Casillas J, Castellino SM, Hudson MM, Mertens AC, Lima IS, Liu Q, Zeltzer LK, Yasui Y, Robison LL, Oeffinger KC. Impact of insurance type on survivor-focused and general preventive health care utilization in adult survivors of childhood cancer: the Childhood Cancer Survivor Study (CCSS). Cancer. 2011 May 1;117(9):1966-75. doi: 10.1002/cncr.25688. Epub 2010 Nov 10. PMID 21509774
- [Background] Keegan TH, Tao L, DeRouen MC, Wu XC, Prasad P, Lynch CF, Shnorhavorian M, Zebrack BJ, Chu R, Harlan LC, Smith AW, Parsons HM; AYA HOPE Study Collaborative Group. Medical care in adolescents and young adult cancer survivors: what are the biggest access-related barriers? J Cancer Surviv. 2014 Jun;8(2):282-92. doi: 10.1007/s11764-013-0332-4. Epub 2014 Jan 10. PMID 24408440
- [Background] Kirchhoff AC, Lyles CR, Fluchel M, Wright J, Leisenring W. Limitations in health care access and utilization among long-term survivors of adolescent and young adult cancer. Cancer. 2012 Dec 1;118(23):5964-72. doi: 10.1002/cncr.27537. Epub 2012 Sep 24. PMID 23007632
- [Background] Mulrooney DA, Yeazel MW, Kawashima T, Mertens AC, Mitby P, Stovall M, Donaldson SS, Green DM, Sklar CA, Robison LL, Leisenring WM. Cardiac outcomes in a cohort of adult survivors of childhood and adolescent cancer: retrospective analysis of the Childhood Cancer Survivor Study cohort. BMJ. 2009 Dec 8;339:b4606. doi: 10.1136/bmj.b4606. PMID 19996459
- [Background] Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res. 2011 May;45(5):626-9. doi: 10.1016/j.jpsychires.2010.10.008. Epub 2010 Oct 28. PMID 21035130

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Navigation Intervention | Enhanced Usual Care
Started | 41 | 41
Completed | 37 | 40
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Population: All participants who consented and completed the baseline survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | Navigation Intervention | Enhanced Usual Care | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 41 | 82
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 44
  Male | 21 | 17 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Pacific Islander | 0 | 2 | 2
  Black | 3 | 2 | 5
  Hispanic | 2 | 2 | 4
  Non Hispanic White | 36 | 35 | 71
Region of Enrollment [Number; unit: participants]
  United States | 41 | 41 | 82

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of the Health Insurance Navigation Program
Description: 10-point (1-10; 1= least helpful and 10= most helpful) scale rating of program quality, including the following (higher scores indicate higher levels of acceptability)-
  * program materials
  * scheduling
  * communication with navigator
  * length and number of sessions (investigator created scale)
Time Frame: 5 month follow-up
Population: The EUC did not complete acceptability measures as it was intended only for the intervention group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Navigation Intervention | Enhanced Usual Care
Number analyzed (Participants) | 37 | 0
units on a scale | 8.9 (1.2) |

2. Primary Outcome: Percentage of Participants Completing All 4 Intervention Sessions
Description: Program feasibility is measured by the percentage of participants completing all 4 intervention sessions.
Time Frame: 1-2 months follow-up
Population: The EUC did not complete any intervention sessions. The percent below reflects % of intervention participants completing all 4 intervention sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | Navigation Intervention | Enhanced Usual Care
Number analyzed (Participants) | 41 | 0
Participants | 33 |

3. Secondary Outcome: Change From Baseline Familiarity With ACA Provisions to 5-month Follow-up
Description: 6 items rating familiarity with key Affordable Care Act (ACA) protections (scores range from 0-6; higher scores indicate higher degree of familiarity) (scale adapted from CCSS Health Insurance Survey)
Time Frame: baseline and 5 month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Navigation Intervention | Enhanced Usual Care
Number analyzed (Participants) | 37 | 40
units on a scale | 1.7 (1.7) | 0.5 (1.6)

4. Secondary Outcome: Change From Baseline Health Insurance Literacy to 5-month Follow-up
Description: 16 items with a 4-category Likert scale ranging from 16-64 (higher scores denoting lower literacy) of confidence on understanding of health insurance terms (higher scores indicate higher levels of health insurance literacy). We report mean health insurance literacy change from baseline to follow-up. Scale adapted from the Urban Institute Health Reform Monitoring Survey-
  * premium
  * deductible
  * co-payments
  * co-insurance
Time Frame: baseline and 5 month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Navigation Intervention | Enhanced Usual Care
Number analyzed (Participants) | 37 | 40
units on a scale | 9.1 (7.6) | 1.8 (7.9)

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Navigation Intervention | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT04520061/Prot_SAP_000.pdf